CLINICAL TRIAL: NCT01408043
Title: A Study of Hematopoietic Stem Cell Supermobilization in Patients With Non-Hodgkin Lymphoma
Brief Title: Etoposide, Filgrastim, and Plerixafor in Improving Stem Cell Mobilization in Treating Patients With Non-Hodgkin Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2410; NCI-2011-01281 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE2410 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-05

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor; Etoposide; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (stem cell supermobilization) (Experimental): Patients receive etoposide IV over 4 hours on day 0, filgrastim SC QD beginning day 1, and plerixafor SC 15-18 hours prior to apheresis. Patients unable to achieve target collection of >= 8 x 10^6 CD34+ cells/kg receive another dose of plerixafor followed by apheresis. Following the second apheresis, patients achieving =< 2 x 10^6 CD34+ cells/kg may continue filgrastim with plerixafor and continue collection according to the attending physician.
  Interventions: Drug: plerixafor; Biological: filgrastim; Drug: etoposide; Procedure: leukapheresis

INTERVENTIONS:
Drug: plerixafor — Given SC
  Other Names: AMD 3100; Mozobil
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Procedure: leukapheresis — Undergo apheresis

SUMMARY:
This clinical trial studies etoposide, filgrastim and plerixafor in improving stem cell mobilization in patients with non-Hodgkin lymphoma. Giving colony-stimulating factors, such as filgrastim, and plerixafor and etoposide together helps stem cells move from the patient's bone marrow to the blood so they can be collected and stored.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of plerixafor improves the proportion of patients with lymphoma who collect >= 8 x 10^6 cluster of differentiation (CD)34+ cells/kg within two days by 25% compared to the historical estimate of 42% with etoposide and G-CSF (filgrastim).

II. To determine whether patients achieving collection of >= 8 x 10^6 CD34+ cells/kg have a 15% one year survival advantage relative to the historical estimate of 68% among patients mobilizing >= 2 but < 8 x 10^6 CD34+ cells/kg with etoposide and G-CSF.

SECONDARY OBJECTIVES:

I. To demonstrate that patients receiving >= 8 x 10^6 CD34+ cells/kg have more rapid neutrophil and platelet recovery and earlier hospital discharge than those receiving < 8 x 10^6 CD 34+ cells/kg.

II. To compare overall survival and progression-free survival between patients receiving >= 8 x 10^6 CD34+ cells/kg and those receiving < 8 x 10^6 CD34+ cells/kg.

III. To compare number of days of apheresis required to achieve goal, transfusion requirements, hospitalization costs, need for remobilization between groups.

IV. To evaluate whether peripheral CD34+ cell count correlates with graft content of CD34+ cells.

OUTLINE:

Patients receive etoposide intravenously (IV) over 4 hours on day 0, filgrastim subcutaneously (SC) once daily (QD) beginning day 1, and plerixafor SC 15-18 hours prior to apheresis. Patients unable to achieve target collection of >= 8 x 10^6 CD34+ cells/kg receive another dose of plerixafor followed by apheresis. Following the second apheresis, patients achieving =< 2 x 10^6 CD34+ cells/kg may continue filgrastim with plerixafor and continue collection according to the attending physician.

After completion of study treatment, patients are followed up at 28 days and then for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy-confirmed non-Hodgkin lymphoma, of any type
* Must be eligible for autologous transplantation according to institutional guidelines
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Karnofsky performance status of 70 to 100
* Negative for human immunodeficiency virus (HIV)
* prior to the start of mobilization, subjects must have:

  * Absolute neutrophil count of >= 1.2 x 10^9/L
  * Platelet count of >= 100 x 10^9/L
  * Creatinine clearance >= 30 mL/minute
* All patients must be able to comprehend and sign informed consent
* If childbearing potential must either agree to complete abstinence from heterosexual intercourse or effective means of contraception during stem cell mobilization and for at least 3 months following last plerixafor dose; female patients will undergo pregnancy test prior to stem cell mobilization therapy

Exclusion Criteria:

* Have had previous transplants and/or prior mobilization attempts
* Have evidence of progressive non-Hodgkin lymphoma
* Have evidence of bone marrow involvement of lymphoma at time of transplant staging
* Had evidence of active central nervous system (CNS) involvement
* Have had previous radiation of the pelvic area
* Have had prior radioimmunotherapy
* Have received experimental therapy within 2 weeks of enrollment
* Be currently enrolled in another investigational protocol
* Have prior history of other malignancies, excluding basal cell carcinoma or squamous cell carcinoma of the skin

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Navneet Majhail, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Stem Cell Supermobilization)
Started | 25
Completed | 24
Not Completed | 1
Not completed — unable to collect cells | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled and received intervention.
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.48 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Collection Using Plerixafor, Etoposide, and Filgrastim
Description: Number of participants able to collect equal to or more than 8 x 10^6 CD34+ cells/kg with addition of plerixafor to etoposide and filgrastim. These participants are defined as supermobilizers. Participants with less than 8 x 10^6 CD34+ cells/kg are defined as normal mobilizers.
Time Frame: Within 2 days of apheresis
Population: All participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 25
Participants
  Supermobilizers | 7
  Normal Mobilizers | 17
  Non mobilizers | 1

2. Primary Outcome: Progression-free Survival
Description: The number of participants of patients who receive greater than or equal to 8 x 10^6 CD34+ cells/kg following collection with plerixafor, etoposide, and filgrastim and that have progression-free survival at one year
Time Frame: Up to 1 year post-transplant
Population: Number of supermobilizer participants that were able to achieve collection of ≥ 8 x 106 CD34+ cells/kg
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 7
Participants | 7

3. Primary Outcome: Overall Survival
Description: Number of participants who receive greater than or equal to 8 x 10^6 CD34+ cells/kg by 15% following collection with plerixafor, etoposide, and filgrastimstill alive at 1 yr post transplant
Time Frame: Up to 1 year post-transplant
Population: Number of supermobilizer participants that were able to achieve collection of ≥ 8 x 106 CD34+ cells/kg
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 7
Participants | 7

4. Secondary Outcome: Neutrophil Recovery in Super Mobilizers and Normal Mobilizers
Description: Neutrophil recovery in participants receiving greater than or equal to 8 and less than 8 x 10^6 CD34+ cells/kg entered as the mean cell count of super mobilizers and normal mobilizers.
Time Frame: Up to 28 days post treatment
Population: All participants that had some mobilization
Measure: Mean (Standard Deviation); unit: K/ul
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
K/ul
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 10.3 (0.5)
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 10.2 (0.7)

5. Secondary Outcome: Platelet Recovery in Super Mobilizers and Normal Mobilizers
Description: Platelet recovery in participants receiving greater than or equal to 8 and less than 8 x 10^6 CD34+ cells/kg.
Time Frame: Up to 28 days post treatment
Population: All participants that had some mobilization
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
percentage of change
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 20.9 (6.5)
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 19.8 (5.6)

6. Secondary Outcome: Length of Hospital Stay in Super Mobilizers and Normal Mobilizers
Description: Length of hospital stay in participants receiving greater than or equal to 8 and less than 8 x 10^6 CD34+ cells/kg.
Time Frame: Up to 28 days post treatment
Population: All participants that had some mobilization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
days
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 20.7 (0.5)
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 22.5 (5.5)

7. Secondary Outcome: Progression-free Survival in Supermobilizers and Normal Mobilizers
Description: Percentage of participants who were alive and free of progression 1 year after transplant (PFS)
Time Frame: Up to 1 year post-transplant
Population: All participants that had some mobilization
Measure: Number; unit: percent of participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
percent of participants
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 100
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 82

8. Secondary Outcome: Overall Survival in Supermobilizers and Normal Mobilizers
Description: Percentage of participants who were alive 1 year after transplant (OS)
Time Frame: Up to 1 year post-transplant
Population: All participants that had some mobilization
Measure: Number; unit: percent of participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
percent of participants
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 100
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 100

9. Secondary Outcome: Number of Days of Apheresis Required
Description: Number of days of apheresis required to achieve goal in supermobilizers and normal mobilizers
Time Frame: Up to 28 days post treatment
Population: Participants that were mobilized
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
days
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 1.1 (0.4)
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 2.9 (1.1)

10. Secondary Outcome: Number of Transfusion Requirements
Description: Number of transfusions (number of packed red blood cells and platelet transfusions required from day 0 to +28 post-transplant) in supermobilizers and normal mobilizers
Time Frame: Up to 28 days post treatment
Population: Participants that were mobilized
Measure: Mean (Standard Deviation); unit: transfusions
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
transfusions
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 3.7 (2.1)
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 4.4 (2.0)

11. Secondary Outcome: Need for Remobilization
Description: Number of participants that needed remobilization in supermobilizers and normal mobilizers.
  Remobilization can be described as follows:
  The first step for patients undergoing autologous hematopoietic cell transplantation is to mobilize hematopoietic progenitor/stem cells from the bone marrow using G-CSF, plerixafor and/or chemotherapy. This is followed by collection of the cells by apheresis. If sufficient number of progenitor/stem cells cannot be mobilized and then collected by apheresis to proceed with transplantation, it is considered as "mobilization failure". For these patients, mobilization of their hematopoietic progenitor/stem cells is attempted a second time ("remobilization"). The need to do a second 'mobilization' attempt is not ideal.
Time Frame: Up to 28 days post treatment
Population: Participants that were mobilized
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 24
Participants
  Supermobilizers: number analyzed (Participants) | 7
  Supermobilizers | 0
  Normal Mobilizers: number analyzed (Participants) | 17
  Normal Mobilizers | 0

12. Secondary Outcome: Correlation of Peripheral CD34+ Cell Count With Graft Content of CD34+ Cells
Description: Correlation of peripheral CD34+ cell count with graft content of CD34+ cells assessed using Spearman correlation.
Time Frame: Up to 28 days post treatment
Population: No data collected for this outcome due to low accrual
Arm/Group | Treatment (Stem Cell Supermobilization)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year post-transplant
Arm/Group | Treatment (Stem Cell Supermobilization)
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes